CLINICAL TRIAL: NCT06505239
Title: A Randomized, Double-Blind, Placebo-Controlled Crossover Study to Assess the Safety and Efficacy of FSD-F2R6-A-CP in Volunteers in an Induced State of Alcohol Intoxication (METAL-2)
Brief Title: Assessing the Safety and Efficacy of FSD-F2R6-A-CP in Volunteers in an Induced State of Alcohol Intoxication
Acronym: METAL-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quantum Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: FSD-F2R6-002
Record Dates: First submitted 2024-07-03; First posted 2024-07-17 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Acute Alcohol Intoxication
MeSH Terms: conditions — Alcoholic Intoxication

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FSD-F2R6-A-CP (Active Comparator)
  Interventions: Dietary Supplement: FSD-F2R6-A-CP
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: FSD-F2R6-A-CP — FSD-F2R6-A-CP is a unique dietary supplement with natural ingredients, vitamins and minerals that potentially enhances cognition, replenishes cofactors needed for alcohol metabolism and may accelerate alcohol metabolism in the body.
  Arms: FSD-F2R6-A-CP
Dietary Supplement: Placebo — Placebo drink designed to match FSD-F2R6-A-CP in color and taste.
  Arms: Placebo

SUMMARY:
This will be a (2 visit) double-blind, randomized, placebo crossover design clinical study to assess the potential benefits of FSD-F2R6-A-CP versus a placebo by assessing its impact on side effect profiles as well as cognitive abilities, motor abilities, and breath alcohol concentration following ingestion of alcohol followed by the dietary supplement or placebo. This study will enroll healthy men and women.

ELIGIBILITY:
Inclusion Criteria:

* English-literate, non-smoking (> 6 months),
* Men and women aged 25 to 45 years,
* Body mass index (BMI) of 18.5 to 32.0 kg/m2, and weighing between 110 and 220 lbs (50-100 kg).
* Free of the diseases listed in exclusion criteria according to their medical history,
* An ECG value of ≤ 440 msec for males and ≤ 460 msec for females, as measured by an FDA-cleared ECG device (6-lead device, KardiaMobile), administered by the investigator.
* Capable of consuming 4-6 standard drinks for women or 5-7 standard drinks for men on a single occasion without experiencing moderate sedation, vomiting, or aggression, to be eligible for the study. Moderate sedation is defined as the subject must be able to communicate and follow simple directions following the consumption of indicated number of drinks.
* Agree not to get tattoos or body piercings, or receive vaccines during the study period, or 7 days prior to the study period.
* Female subjects who must test negative on a urine pregnancy test, and cannot be pregnant or lactating. All subjects are required to either refrain from sex or use at least one form of contraception throughout the study, including a condom or either an oral or intrauterine contraceptive.
* Men who must agree not to donate sperm for 90 days following the trial.
* Experienced at least 2 hangovers
* Clinical laboratory values within the most recent acceptable laboratory test range, and/or values are deemed by the Investigator /Sub-Investigator as "Not Clinically Significant" as per CBC/CMP, urinalysis, and coagulation testing.

Exclusion Criteria:

* A known history or presence of any clinically relevant conditions affecting the liver, kidneys, gastrointestinal system, cardiovascular system, cerebrovascular system, lungs, endocrine system, immune system, musculoskeletal system, nervous system, psychiatric state, respiratory system, skin, or blood, unless deemed not clinically significant by the Investigator/Sub-Investigator. This includes a significant history or current issues with gastrointestinal pathology, such as chronic diarrhea or inflammatory bowel diseases, or conditions affecting drug absorption, distribution, metabolism, or excretion
* Major surgery within the past 6 months, a history of seizures, significant head trauma, or neurosurgery, or any clinically significant illness within 30 days prior to dosing are also excluded
* Are on a ketogenic or very low carbohydrate diet within the past 30 days.
* Significant physical or organ abnormalities, a positive screening for a HIV, Hepatitis B or C (as determined by medical health questionnaires), or positive test result for drugs with abuse potential (cannabis, amphetamines, barbiturates, cocaine, opiates, phencyclidine and benzodiazepines)
* Alcohol-naïve
* Positive pregnancy test
* A history of significant alcohol sensitivity
* A history of adverse reactions to power (energy) drinks or caffeine,
* Severe food allergies, or dietary restrictions.
* Allergic reactions to any ingredients in the FSD-F2R6-A-CP and placebo.
* A psychiatric history of certain disorders, a first-degree relative with specific psychiatric or alcohol use disorders,
* An intolerance to blood sampling, recent blood or plasma donations within the past 60 days.
* Recently used enzyme-modifying drugs within the previous 30 days including strong inhibitors of cytochrome P450 (CYP) enzymes (e.g., cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and HIV antivirals) and strong inducers of CYP enzymes (e.g., barbiturates, carbamazepine, glucocorticoids, phenytoin, St. John's Wort, and rifampicin).
* Current or past history within the last 2 years of alcohol or drug dependence (excluding caffeine and nicotine).
* Current or past history within the last 5 years of major depressive disorder, obsessive-compulsive disorder, panic disorder, anorexia nervosa, or bulimia nervosa. First-degree relative with current or historical Alcohol Use Disorder (AUD).
* Intolerance to and/or difficulty with blood sampling through venipuncture or indwelling catheter.
* Used of prescription medication (other than contraception or occasional paracetamol) or over-the-counter medications including supplements within 14 days prior to session 1,
* A positive alcohol test at check-in on treatment day,
* Recent tattoos or piercings (within 7 days of study enrollment)
* Any condition deemed by the Investigator or Sponsor to interfere with study participation will be excluded.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2024-07-12 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-11-07 (Actual)

PRIMARY OUTCOMES:
Intoxication | Change in pre-treatment score to 0.5, 1, 2 and 4 hours post-treatment
  Intoxication will be measured using a 0-100 mm VAS scale, with left (0 mm) and right (100 mm) anchors designated 'not at all' and 'very much' to assess subjects' subjective experience of intoxication.
Impairment | Change in pre-treatment score to 0.5, 1, 2 and 4 hours post-treatment
  Impairment will be measured using a 0-100 mm VAS scale, with left (0 mm) and right (100 mm) anchors designated 'not at all' and 'very much' to assess subjects' subjective experience of impairment.
Mental Fatigue | Change in pre-treatment score to 0.5, 1, 2 and4 hours post-treatment
  Mental fatigue will be measured using a 0-100 mm VAS scale, with left (0 mm) and right (100 mm) anchors designated 'not at all' and 'very much' to assess subjects' subjective experience of mental fatigue.
Clearheaded-Muzzy | Change in pre-treatment score to 0.5, 1, 2 and 4 hours post-treatment
  Clearheaded-Muzzy will be measured by a 100 mm visual analog scale (VAS) representing bipolar adjective pairs for the assessment of both alerting and sedating CNS drug effects.
Clumsy-Well Coordinated | Change in pre-treatment score to 0.5, 1, 2 and 4 hours post-treatment
  Clumsy-Well Coordinated will be measured by a 100 mm visual analog scale (VAS) representing bipolar adjective pairs for the assessment of both alerting and sedating CNS drug effects.
Energetic-Lethargic | Change in pre-treatment score to 0.5, 1, 2 an 4 hours post-treatment
  Energetic-Lethargic will be measured by a 100 mm visual analog scale (VAS) representing bipolar adjective pairs for the assessment of both alerting and sedating CNS drug effects.
Drowsy-Alert | Change in pre-treatment score to 0.5, 1, 2 an 4 hours post-treatment
  Drowsy-Alert will be measured by a 100 mm visual analog scale (VAS) representing bipolar adjective pairs for the assessment of both alerting and sedating CNS drug effects.
Mentally Slow-Quick Witted | Change in pre-treatment score to 0.5, 1, 2 and 4 hours post-treatment
  Mentally Slow-Quick Witted will be measured by a 100 mm visual analog scale (VAS) representing bipolar adjective pairs for the assessment of both alerting and sedating CNS drug effects.
Headache | Change in pre-treatment score to 0.5, 1, 2, 4 and 8 hours post-treatment
  Headache will be measured on a 100 mm VAS. The subject will indicate the severity of any headache by drawing a vertical line on the horizontally positioned VAS. The left end (0 mm) of the VAS will designate 'no pain' and the right end (100mm) will designate 'most severe pain imaginable' with no intermediate divisions or descriptive terms.

SECONDARY OUTCOMES:
Druid App Test | Change in pre-treatment score to 0.5, 1, 2 and 4 hours post-treatment
  This is a peer-reviewed, phone app with 4 different tests that test for cognitive and motor impairments.
Digital Symbol Substitution Task (DSST) | Change in pre-treatment score to 0.5, 1, 2 and 4 hours post-treatment
  This is a computerized test that will be used to assess the subject's cognitive functioning. This will test processing speed, working memory, visuospatial processing and attention.
Trail Making Test (TMT) | Change in pre-treatment score to 0.5, 1, 2 and 4 hours post-treatment
  This is a neuropsychological test of visual attention and task switching. Subjects will connect a set of 25 dots in order as quickly and accurately as possible. This will provide visual search speed, scanning, speed of processing, mental flexibility, and executive functioning. This test will be completed on a computer.
Breath Alcohol Concentration | Change in pre-treatment score to 0.5, 1, 1.5, 2, 3 and 4 hours post-treatment
  To quantify the participants' level of intoxication through objective measures, breath alcohol concentrations will be measured with a breathalyzer.
Acute Hangover Severity Scale (AHSS) | Measured at 8 and 24 hours after treatment
  This is a 12-item questionnaire that rates the severity of a hangover from 0 to 120 with higher scores indicating worse hangover symptoms.
Single Item Hangover Severity Score | Measured at 8 and 24 hours after treatment
  This is a single item outcome measure that rates the severity of a hangover from 0 to 10 with higher scores indicating worse hangover symptoms.
Systolic blood pressure | Measured at baseline (before alcohol), pre-treatment and 0.5, 1, 2 and 4 hours post-treatment
  Systolic blood pressure measured in mmHg.
Diastolic blood pressure | Measured at baseline (before alcohol), pre-treatment and 0.5, 1, 2 and 4 hours post-treatment
  Diastolic blood pressure measured in mmHg
Heart rate | Measured at baseline (before alcohol), pre-treatment and 0.5, 1, 2 and 4 hours post-treatment
  Heart rate measured in beats per minute
Respiratory rate | Measured at baseline (before alcohol), pre-treatment and 0.5, 1, 2 and 4 hours post-treatment
  Respiratory rate measured in respirations per minute
Temperature | Measured at baseline (before alcohol), pre-treatment and 0.5, 1, 2 and 4 hours post-treatment
  Temperature measured in degrees fahrenheit with an infrared thermometer

OTHER OUTCOMES:
Adverse Events (AEs) | Pre-treatment until 24 hour post-treatment visit
  Incidence of AEs will be determined based on observation and verbal subject questioning.
Complete blood count (CBC) | Change in test results from baseline to 24 hours post-treatment
  Safety blood test measured by a laboratory using a reference range
Comprehensive metabolic blood panel (CMP) | Change in test results from baseline to 24 hours post-treatment
  Safety blood test measured by a laboratory using a reference range
Blood coagulation | Change in test results from baseline to 24 hours post-treatment
  Safety blood test measured by a laboratory using a reference range

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sikorski, PhD, Principal Investigator — Applied Science and Performance Institute
Locations (1):
- Applied Science and Performance Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No